CLINICAL TRIAL: NCT06550778
Title: Ethics Committee of Daqing Campus of Harbin Medical University
Brief Title: Construction and Preliminary Application of Mindfulness-based Emotional Regulation Intervention Scheme for Adolescents With Anxiety Disorder and Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhan Yuxin (Other)
Responsible Party: Sponsor-Investigator, Zhan Yuxin, researcher, Harbin Medical University
Organization: Harbin Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HMUDQ20230913001
Record Dates: First submitted 2024-08-07; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Anxiety; Mindfulness; Emotional Regulation
MeSH Terms: conditions — Anxiety Disorders; Emotional Regulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: Mindfulness-based emotional regulation intervention
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Mindfulness-based emotional regulation intervention — The intervention was conducted once a week for 6 weeks, with each session lasting 90-120 minutes, including a 30-minute parenting course each week. The intervention program was divided into 6 themes, including "Entering mindfulness, feeling the connection between emotions and the body", "Dealing with negative emotions", "Moderate emotional expression", "Mindfulness to relieve anxiety", "Learning to be grateful" and "Embrace future life". The intervention content integrates mindfulness training, parental mindful parenting exercises and emotion regulation skills. For details, refer to Greenland's "Mindfulness Games", Bögels' "Mindful Parenting Manual", mindful breathing and meditation in MBSR and MBCT, as well as emotion regulation skills. The intervention location was the activity room of the child and adolescent psychology unit of the hospital.
  Arms: Intervention group

SUMMARY:
Purpose：Aiming to improve the emotional regulation abilities of adolescents with AD and caregivers, reduce anxiety levels, and play an important role in promoting the recovery of adolescents with AD and the mental and physical health of parents.

Methods：This study is divided into two parts. In Part One, a mindfulness-based emotional regulation intervention program for adolescents with anxiety disorders and their caregivers was developed. Drawing on family systems theory, the mindfulness coping model, and Gross's emotion regulation process model, a systematic literature review was conducted to extract the main contents of the intervention program. Semi-structured interviews were conducted with 11 pairs of adolescents with AD and their caregivers to identify emotional regulation issues and intervention needs, forming a preliminary draft of the mindfulness-based emotional regulation intervention program for adolescents with anxiety disorders and their caregivers. Fifteen experts were invited to participate in Delphi consultations, and based on pre-experimental feedback, the intervention program was further refined to produce a pilot intervention protocol.

In Part Two, the feasibility and effectiveness of the mindfulness-based emotional regulation intervention for adolescents with anxiety disorders and their caregivers were preliminarily assessed. Using a randomized controlled trial design, 78 pairs of adolescents with AD and their caregivers who met the inclusion criteria were selected from the Children and Adolescent Psychological Unit at the Third Hospital of Daqing City, Heilongjiang Province. They were randomly assigned to either the intervention group (n=39 pairs) receiving a 6-week mindfulness-based emotional regulation intervention or the control group (n=39 pairs) receiving routine hospital care. During the intervention period, 4 adolescents with AD and 5 caregivers withdrew from the intervention group, while 2 adolescents with AD and 3 caregivers withdrew from the control group. Assessments were conducted at baseline (T0), immediately post-intervention (T1), and one month post-intervention (T2) using the Emotion Regulation Questionnaire (ERQ), Self-Rating Anxiety Scale, Mindful Attention Awareness Scale (MAAS), Ruminative Responses Scale (RRS), and Mindfulness in Parenting Questionnaire (MIPQ) for both adolescents with AD and their caregivers. Data were analyzed using SPSS 26.0, employing descriptive statistics, t-tests, chi-square tests, Mann-Whitney U tests, and generalized estimating equations to compare the intervention effects.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents aged 12-18 years who meet the diagnostic criteria of the 10th edition of the International Classification of Diseases (ICD-10) and are diagnosed with AD by clinical psychiatrists and have a score of ≥50 on the anxiety self-rating scale;
2. Adolescents are treated with benzodiazepines or 5-HT reuptake inhibitors;
3. Adolescents are in stable condition and have been hospitalized for at least 6 weeks;
4. Adolescents can communicate normally and voluntarily participate in this study;
5. The father or mother of the AD adolescent who meets the above inclusion criteria;
6. As the main fixed caregiver of the child, they are mainly responsible for daily care work, taking care of the child for ≥5 days per week and taking care of the child for more than 3 months ;
7. Informed consent and voluntarily participate in this study.

Exclusion Criteria:

1. The caregiver has severe cognitive impairment, mental illness, and physical illness;
2. The AD adolescent and the caregiver have participated in other psychological interventions or researchers within 6 months;
3. The AD adolescent cannot continue to cooperate with the study due to worsening of the condition;
4. Voluntarily withdraw from the study midway.

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 78 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Emotion Regulation Questionnaire | 10weeks
  The questionnaire was compiled by Gross and John et al. in 2003 and is used to evaluate the level of emotion regulation. This study used the Chinese version translated by Wang Li et al. [142]. The questionnaire contains two dimensions, namely cognitive reappraisal and expressive inhibition, with a total of 10 items, and is scored on a scale of 1-7 (1 = "strongly agree", 7 = "strongly disagree"). The Cronbach's α coefficient for the cognitive reappraisal dimension of the questionnaire is 0.85, and the Cronbach's α coefficient for the expressive inhibition dimension is 0.77; in this study, the Cronbach's α coefficient for the cognitive reappraisal dimension is 0.83, and the Cronbach's α coefficient for the expressive inhibition dimension is 0.79.
Self-rating Anxiety Scale | 10weeks
  The scale was compiled by foreign scholar Zung in 1971. It aims to objectively reflect the patient's subjective emotions and assess the degree of anxiety symptoms. The scale contains 20 items, which are scored on a 1-4 scale (1 = "never or rarely"; 4 = "most or all of the time"). The standard score is the total score * 1.25, and the sum of the scores of the 20 items is the total score. A standard score ≥ 50 indicates anxiety symptoms. In this study, the Cronbach's α coefficient was 0.87.

SECONDARY OUTCOMES:
Mindful Attention Awareness Scale | 10weeks
  The questionnaire was developed by Brown and Ryan in 2003. It is used to assess people's perception of their daily life experiences, mainly including cognitive, emotional and physiological aspects. This study used the Chinese version of the Mindfulness Awareness Scale revised by Chen Siyi, Cui Hong, Zhou Renlai and Jia Yanyan [143]. The scale has 15 items, which are scored on a scale of 1-6 (1 = "never", 6 = "always"). The total score of the scale ranges from 15 to 90. The scoring standard is: the higher the total score of the scale, the higher the degree of mindfulness of the subject. MAAS has good internal consistency, with a Cronbach's α coefficient of 0.85 . In this study, the Cronbach's α coefficient was 0.87.
Ruminative Responses Scale | 10weeks
  The Ruminative Responses Scale (RRS) was developed by Nolen-Hoeksema in 1991. The scale was revised by Han Xiu and Yang Hongfei to form the Chinese version of the ruminative thinking scale [144]. The scale has 22 items, including three dimensions: symptom rumination, obsessive thinking, and reflective thinking. It is scored on a 1-4 scale (1 = "never", 4 = "always"), and the higher the score, the more severe the tendency of rumination. The Cronbach's α coefficient of the scale is 0.90 , and the Cronbach's α coefficient in this study is 0.88.
Mindfulness in Parenting Questionnaire | 10weeks
  The Mindfulness in Parenting Questionnaire (MIPQ) was developed by McCaffrey and revised in Chinese by Zhao Yaping et al. It includes two dimensions: focusing on the present and mindful parenting. It has 28 items and is scored on a 1-4 scale (1 = "occasionally", 4 = "always"). The higher the individual's mindful parenting behavior, the higher the final score. Cronbach's α coefficient is 0.90 [144]. In this study, Cronbach's α coefficient was 0.86.

CONTACTS AND LOCATIONS:
Locations (1):
- Harbin Medical University, Daqing, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No